CLINICAL TRIAL: NCT01654055
Title: International Multicentre Prospective Study on Morphine-induced Adverse Drug Reactions in Emergency Departments: Description and Predictive Factors.
Brief Title: International Prospective Study on Morphine-induced Adverse Drug Reactions in Emergency Departments.
Acronym: EI-Morphinique
Status: Completed | Type: Observational
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: 1243803
Record Dates: First submitted 2012-07-27; First posted 2012-07-31 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Emergencies
Keywords: Morphine; Adverse events; Predictive factors
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Morphine is the gold standard for treatment of severe acute pain but it has a number of adverse effects.

No study has so far managed to identify the morphine-induced adverse drug reactions. The primary objective of this study is to determine predictive factors of morphine-induced adverse drug reaction when it is used in emergency departments.

DETAILED DESCRIPTION:
We want to study a large cohort of morphine-induced adverse drug reactions patients, the consequences for patients, mainly in terms of severity, and predictive criteria. This will allow us to identify some patients most at risk of morphine-induced adverse drug reactions, and thus to adapt morphine titration and monitoring of these patients. Leading to a better understanding and a better prediction of adverse effects in patients, it is possible that part of the "opiophobia" which persists in emergency services disappear. Finally, it is toward a better security but also a better efficiency in the management of pain patients in emergencies that leads this study.

The secondary objectives are:

To determine the frequency and severity of adverse events related to morphine. To establish an inventory of morphine use in emergency departments in the different centres studied.

ELIGIBILITY:
Inclusion Criteria:

All patients aged 18 years or older who require treatment with morphine for pain control will be considered for entry into the study.

Conscious without life threatening at the inclusion

Exclusion Criteria:

Patients who receive morphine during or after an orotracheal intubation, altered level of consciousness, inability to give consent or refusal of patient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 18 years or older who require treatment with morphine for pain control
Sampling Method: Probability Sample
Enrollment: 1128 (Actual)
Dates: Start 2011-10; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Occurrence of morphine related adverse-event | From the administration of morphine until 6 hours after this first administration
  The primary outcome variable will be defined as occurrence of morphine related adverse-event (including nausea, dizziness, emesis, drowsiness, pruritus, respiratory distress and death)

SECONDARY OUTCOMES:
Description of adverse effects caused by morphine | For each side effects of morphine from the first administration of morphine until 6 hours after.
  Description of adverse effects caused by morphine, initial and final pain scores and support given by centres. Imputability scores will be evaluated for each event.

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Bounes, MD, Principal Investigator
Locations (1):
- University Hospital Toulouse, Toulouse, Midi-Pyrénées, France

IPD SHARING:
Plan to Share IPD: No